CLINICAL TRIAL: NCT05594823
Title: Flexible vs. Fixed Diuretic Regimen in the Management of Chronic Heart Failure: A Pilot Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Stuart Smith, MD, Cardiologist, Director of Heart Failure Services, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDA ID: 12724
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Heart Diseases
Keywords: diuretic; furosemide; flexible diuretic regimen; weight-based
MeSH Terms: conditions — Heart Failure; Heart Diseases | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fixed - dose diuretic (Active Comparator): Pre-determined, fixed daily dose of diuretic (furosemide)
  Interventions: Other: Ambulatory heart failure management with fixed dose furosemide
- Flexible diuretic regimen (Experimental): Variable daily dose of diuretic (furosemide) determined based on a pre-specified weight-based scale.
  Interventions: Other: Ambulatory heart failure management with Flexible Diuretic Regimen with furosemide

INTERVENTIONS:
Other: Ambulatory heart failure management with Flexible Diuretic Regimen with furosemide — Subjects will be given a regimen that determines a variable daily dose of diuretic (furosemide) based on daily self-measured weights as part of the standard of care ambulatory management of chronic heart failure. Follow-up will occur at 90 days with routine bloodwork to monitor renal function.
  Arms: Flexible diuretic regimen
Other: Ambulatory heart failure management with fixed dose furosemide — Subjects will be prescribed a fixed daily dose of diuretic (furosemide) as part of the standard of care ambulatory management of chronic heart failure. Follow-up will occur at 90 days with routine bloodwork to monitor renal function.
  Arms: Fixed - dose diuretic

SUMMARY:
Heart failure is a major cause of death and hospitalization in Canada. Many of the symptoms experienced by patients with heart failure relate to having fluid accumulate in the lungs causing difficulty breathing, swelling in the legs, and an increase in weight. Thus, one of the cornerstones of managing heart failure includes the use of medications known as diuretics that target the kidneys to reduce fluid accumulation via urination. Deciding on the correct dose of this medication can be quite nuanced as under-dosing can lead to accumulation of fluid, and over-dosing can dehydrate patients and potentially result in lightheadedness/fainting and damage to the kidneys. Currently, options for prescribing diuretics for heart failure include 1) giving patients a regular, fixed dose or 2) having patients monitor their daily weight as a surrogate of their fluid status and then take a dose of diuretic based on a pre-prepared scale. The rationale behind the flexible weight-based diuretic scale is that it can potentially detect early fluid accumulation and thus possibly prevent hospitalization or ED visits, and it also avoids over-dosing and potentially dehydrating patients. Currently, it is not clear whether the flexible diuretic regimen is better than the fixed-dose regimen in preventing ED visits, hospitalizations, kidney damage, or death and as such, this pilot study will directly compare the two commonly used regimens in the management of chronic heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of heart failure, either reduced (Left ventricular ejection fraction [LVEF] ≤ 40%) or preserved (LVEF > 40%) ejection fraction as measured by echocardiography performed within the last 2 months
2. Prescribed and tolerating furosemide with a minimum daily dose of 40mg oral daily
3. New York Heart Association (NYHA) Class II or higher symptoms
4. NT-proBNP cutoff of ≥ 1000 pg/mL performed within 30 days prior to randomization
5. Age > 18 years
6. English speaking
7. Access to a scale and ability to weigh themselves daily and reliable telephone access

Exclusion Criteria:

1. Myocardial infarction, coronary artery bypass graft surgery, stent insertion and/or angioplasty within 14 days
2. Pregnancy
3. Inability to follow directions and self-monitor as part of a flexible diuretic regimen as discerned by the clinician
4. Allergic reaction to loop diuretics
5. Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Mortality and morbidity composite outcome | 90 days
  Time to first event of a composite outcome including: ambulatory heart failure visit (clinic or emergency department) requiring intravenous diuretic, an increase in oral diuretic dose greater than or equal to 2.5 times their baseline dose prescribed at time of randomization, or the addition of metolazone; hospitalization for heart failure and/or acute kidney injury defined as a serum creatinine > 1.5 times from baseline at time of randomization; and all-cause death up to 90 days post-randomization

SECONDARY OUTCOMES:
Incidence of acute kidney injury | 90 days
  Rate of acute kidney injury defined as a serum creatinine increase of >1.5 times from baseline at 90 days from randomization
Heart Failure Hospitalizations | 90 days
  Total number of hospitalizations due to heart failure (first and recurrent) during the 90 days post-randomization
All-cause Hospitalizations | 90 days
  Total number of hospitalizations for any cause during the 90 days post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Smith, MD, Principal Investigator — Western University
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No